CLINICAL TRIAL: NCT06902675
Title: Artificial Intelligence as a Decision Making Tool in Neurology
Status: Active, not recruiting | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, . Shahr Shelly MD, Specialist in Neurology and Immunology, Rambam Health Care Campus
Other Study IDs: 0026-24RMB
Record Dates: First submitted 2024-11-13; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Clinical Decision-making; Medical Reporting; Neurological Diseases or Conditions; Emergency Department Visit
MeSH Terms: interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Evaluation With AI: * Description: Participants in this arm receive an LLM-based recommendation that is presented to the resident (after senior physician approval) given by random selection (control versus study) 1:1.
  * Intervention: Artificial Intelligence as a Decision-Making Tool
  * Intervention Description: The large language model (LLM) provides clinical suggestions regarding diagnosis or management. The final decision remains at the discretion of the attending physician.
  Interventions: Other: Artificial Intelligence
- Evaluation Without AI: * Description: Participants in this arm receive standard clinical care without access to an AI-based recommendation given by random selection (control versus study) 1:1 to the neurological resident.
  * Intervention: No Intervention
  * Intervention Description: Standard of care only. No AI tool is provided to the resident.
- Retrospective Cohort: * Description: Clinical data from 10,000 patients previously evaluated by neurologists in the Emergency Department are extracted and analyzed retrospectively.
  * Intervention: Data Extraction and Analysis
  * Intervention Description: De-identified data are uploaded into the LLM for retrospective analysis. Model outputs are then compared to actual patient outcomes and standard-of-care decisions.
  Interventions: Other: Retrospective Data Extraction of 10,000 Neurology ER Cases

INTERVENTIONS:
Other: Artificial Intelligence — Artificial Intelligence as a decision making tool
  Groups: Evaluation With AI
Other: Retrospective Data Extraction of 10,000 Neurology ER Cases — This intervention involves collecting and de-identifying clinical data from 10,000 patients previously evaluated by neurologists in the Emergency Department. The data are then used retrospectively to refine and fine-tune a large language model (LLM). No real-time clinical decisions or recommendations are made for these patients, as the purpose is to improve the model's accuracy and relevance for future use.
  Groups: Retrospective Cohort

SUMMARY:
Background: The establishment of neuroinformatics as a distinct field has enabled the integration of computational biology and informatics to improve neurological research. This interdisciplinary approach enhances the capacity to integrate diverse datasets, unravel complex neural networks, and develop computational models that can improve clinical management. The investigators aim to evaluate whether an artificial-intelligence-based tool is effective in non-English-speaking regions.

Hypothesis: Integrating a language model-based clinical assistance system within the neurology ward will significantly enhance the efficiency and accuracy of patient care by leveraging neuroinformatics principles. The investigators hypothesize that combining natural language processing and data analytics will improve diagnostic and treatment processes.

DETAILED DESCRIPTION:
Research Design:

A pre-post-intervention design will be used, measuring outcomes before and after the implementation of a neuroinformatics-driven clinical assistance system. Changes in diagnostic accuracy, treatment decisions, and workflow efficiency will be quantified.

Workflow:

1. A neurologist evaluates each patient, and the patient signs informed consent.
2. A medical student manually uploads de-identified clinical information to a secure interface.
3. Data are analyzed by a large language model (LLM) system through a hospital-approved application.
4. A senior physician must approve any decision based on the LLM's recommendation.
5. For half of the prospectively enrolled participants, the LLM's recommendation is presented to the resident.

Retrospective Data:

1. The investigators will extract data from 10,000 patients who were evaluated by a neurologist in the Emergency Department.
2. Clinical information (without patient identifiers) will be uploaded to a secure, hospital-approved LLM with a security key.
3. The model's output will be compared with actual clinical decisions and patient outcomes (e.g., mortality, discharge status).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent

Exclusion Criteria:

* Unable to give informed consent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥18 years) receiving care in Neurology Department A, including both patients hospitalized in the neurological ward (Department A) and outpatients from the neurology department's clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of correct diagnoses generated by the LLM compared to the final attending physician diagnosis. | 3 years
  * Description: Measures the percentage of times the LLM's recommended diagnosis matches the final attending physician's diagnosis.
  * Unit of Measure: Proportion (0.0-1.0) or Percent (0-100%)
  * How Assessed: Each LLM recommendation is compared to the final documented diagnosis in the medical record. The number of correct diagnoses is divided by the total number of cases.
Accuracy of Next-Step Recommendations | Up to 3 years.
  Proportion of correct or appropriate next-step management decisions recommended by the LLM.
  Description: Proportion of correct next-step management decisions recommended by the LLM, compared to either the attending physician's final plan or standard-of-care guidelines.
  Unit of Measure: Proportion (0.0-1.0) or Percent (0-100%) How Assessed: For each encounter, the LLM's recommended "next step" is recorded and deemed correct if it aligns with the attending plan or guideline.

SECONDARY OUTCOMES:
Cost of Running the LLM | Up to 3 years
  Average daily cost (in USD) to operate the large language model.
  Description:
  This outcome will measure the direct computational and licensing costs incurred by running the LLM in the clinical setting.
  Unit of Measure: US Dollars (per day). How It Is Assessed: The total daily spend for the LLM (e.g., cloud-compute fees, licensing fees) will be recorded and divided by the total number of patient encounters that day to derive an average cost.
Staff Compliance With AI | Up to 3 years
  This outcome will assess how often (compliance) and how willingly (acceptance) physicians, residents, and nurses use the LLM in eligible clinical scenarios.
  Description: Determines how often physicians, residents, and nurses use the LLM for eligible patient encounters.
  Unit of Measure: Proportion (0.0-1.0) or Percent (0-100%) How Assessed: Tracks the number of encounters in which the LLM is actually used, divided by the total number of eligible encounters. Higher percentages indicate greater compliance.
Transparency/Explainability | 3 years
  Description: Evaluates how clearly the LLM's reasoning is communicated to clinical staff.
  Unit of Measure: Score on a 5-point Likert scale (1 = not at all clear, 5 = extremely clear) How Assessed: After each LLM-guided decision, the resident or attending physician rates the clarity of the model's explanation. A mean score is reported. Higher scores indicate better clarity.
Quality of LLM-Generated Clinical Reports | Up to 3 years
  Accuracy and Completeness Score of the LLM-Generated Clinical Report This outcome evaluates how accurately and comprehensively the LLM summarizes a patient's clinical encounter and recommended plan in a structured report (e.g., discharge instructions, progress notes).
  Unit(s) of Measure: Quality Score based on a modified SOAP (Subjective, Objective, Assessment, Plan) Note Rating Scale, ranging from 0 to 10, where higher scores indicate better documentation quality. The score reflects the inclusion of required elements and correctness of clinical details.
  Assessment Method: Each LLM-generated report is independently evaluated by a panel of attending physicians or trained clinical staff. Using a standardized checklist, reviewers assess completeness (e.g., inclusion of symptoms, physical findings, diagnosis, and plan) and accuracy (e.g., correct medications, identifiers, and diagnoses), then assign a score based on the predefined rubric.
Staff Acceptance of AI | Up to 3 years
  Description: Evaluates how willingly staff integrate the LLM into their clinical workflow.
  Unit of Measure: 5-point Likert scale (1 = strongly disagree, 5 = strongly agree) How Assessed: After each LLM-assisted encounter, staff complete a brief survey about perceived helpfulness and willingness to reuse the LLM. Higher scores indicate greater acceptance.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam healthcare campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorenshtein A, Weisblat Y, Khateb M, Kenan G, Tsirkin I, Fayn G, Geller S, Shelly S. AI-Based EMG Reporting: A Randomized Controlled Trial. J Neurol. 2025 Aug 22;272(9):586. doi: 10.1007/s00415-025-13261-3. PMID 40844612